CLINICAL TRIAL: NCT01219257
Title: Longitudinal ULtrasonographic Study of Patients With Spondylarthritis Starting First Time or Switching to a New Biological Therapy; the ULSpABiT Study.
Brief Title: Longitudinal ULtrasonographic Study of Patients With Spondylarthritis Starting Biological Therapy
Acronym: ULSPABIT
Status: Completed | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Hilde Berner Hammer, Senior consultant, PhD, Diakonhjemmet Hospital
Other Study IDs: 011110
Record Dates: First submitted 2010-09-15; First posted 2010-10-13 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Spondyloarthritis; Ultrasonography
Keywords: SpA; Anti-TNF alpha treatment; Ultrasonography; Synovitis; Enthesitis
MeSH Terms: conditions — Spondylarthritis; Synovitis | interventions — Adalimumab; Etanercept; Infliximab; golimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the first visit, one glass with blood will be frozen for later genetical analyzes, all related to questions regarding SpA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SpA patients: The patients may be included when their rheumatologist has decided that the patient are going to start biological medication.
  Interventions: Biological: Anti-TNF alpha therapy

INTERVENTIONS:
Biological: Anti-TNF alpha therapy — All medical treatment will be standardizes following good medical practice
  Other Names: Adalimumab (HumiraR); Etanercept (EnbrelR); Infliximab (RemicadeR); Golimumab (SimponiR)

SUMMARY:
Patients with spondylarthritis (SpA) (including ankylosing spondylitis, psoriatic arthritis, arthritis as part of inflammatory bowel disease and reactive arthritis) have axial involvement (the spine) as well as peripheral inflammation in joints and entheses (where the tendons and ligaments are anchored to the bone). Patients with high disease activity of SpA may need biological treatment (anti-TNF alpha), which are very expensive medications. Thus it is necessary to have a sensitive method for assessing the response to treatment. Ultrasonography (US) is a validated and reliable method for assessing disease activity in joints and tendons, and may be used to follow the treatment response.

The present study will include patients with SpA starting on anti-TNF alpha treatment (as first biologic medication or when switching to a new biologic treatment). The study is an extension of the ongoing NORDMARD study (Norwegian longitudinal observational study of arthritic patients starting disease-modifying treatment). The patients will be examined by use of US of 38 joints and 14 entheses at baseline and after 3, 6 and 12 months.

The objectives are to explore US as a method to assess peripheral inflammatory activity for evaluation of response to medication as well as to compare the US pathology with clinical and laboratory findings.

ELIGIBILITY:
Inclusion Criteria:

* SpA
* Planning to start anti-TNF alpha treatment

Exclusion Criteria:

* Patients not being able to communicate in Norwegian or not being able to fill in questionnaires
* Surgery in more than 5 of the joints/entheses to be examined by US

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SpA patients with high disease activity
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To assess the sensitivity to change of US pathology in joints and entheses in SpA patients starting biological treatment. | Including patients for about 1.5 years
  The joints will be assessed according to a US atlas by use of a semi-quantitative (0-3) scoring system and the entheses will be evaluated according to internationally accepted scoring methods.

SECONDARY OUTCOMES:
1. Explore whether the US (B-mode and power Doppler) scores at baseline or after 3 months predict patients responding to biological treatment after 6 and 12 months. | 2.5 years
2. Explore whether the sensitivity for change is higher for US (B-mode and/or power Doppler) than for the traditional assessments for inflammatory activity. | 2.5 years
3. Explore potential differences of US detected pathology in joints and entheses between subgroups of spondylarthritis patients. | 2.5 years
4. Explore whether the different subgroups of spondylarthritis patients have different US response (B-mode synovitis and power Doppler in joints and entheses) to biological treatment. | 2.5 years
5. Explore the association between the US findings (BM and/or PD) and the patient's experience of pain and fatigue. | 2.5 years
6. Explore the associations between calprotectin and US detected inflammation in joints and/or entheses as well as traditional assessments of disease activity. | 2.5 years
  Calprotectin, a major granulocyte protein, is assessed by use of ELISA in plasma. Plasma samples will be frozen at all visits, and the calprotectin assessments will be performed when all patients have finished the study.
7. Explore whether baseline calprotectin or other biomarkers in blood may predict response to biological medication. | 2.5 years
  Plasma and serum will be frozen at each visit, and the S100 proteins calprotectin as well as A12 will be assessed. In addition, other relevant biomarkers may be analyzed after 2.5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde B Hammer, MD, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Department of Rheumatology, Diakonhjemmet Hospital, Oslo, Norway